CLINICAL TRIAL: NCT01108939
Title: The Effect of Asymptomatic Malaria on Iron Absorption and Utilization From a Sorghum-based Meal in Adult Women in Benin
Brief Title: Study of Iron Absorption and Utilization in Asymptomatic Malaria
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof., Swiss Federal Institute of Technology
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Fe_Malaria_Benin
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Malaria, Falciparum
Keywords: Malaria, Iron absorption, Iron utilization, Benin
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antimalarial treatment (Experimental)
  Interventions: Drug: Antimalarial treatment
- Observation (Sham Comparator)
  Interventions: Other: Observation

INTERVENTIONS:
Drug: Antimalarial treatment
  Arms: Antimalarial treatment
Other: Observation
  Arms: Observation

SUMMARY:
Anemia is still a main public health problem in sub-Saharan Africa. Anemic women have an increased maternal and perinatal mortality and anemic adults have diminished work capacity. In sub-Saharan Africa, the etiology of anemia is multifactoral; the major causes are low dietary bioavailability and chronic parasitic infections such as malaria. These causes are likely to interact because infection and infection-associated inflammation may impair the utilization and absorption of iron. Therefore, the control of parasite infections may be important to improve iron bioavailability from foods.

Malaria infections are endemic in northern Benin. To investigate the contribution of asymptomatic malaria (a positive blood smear for malarial parasites but without clinical symptoms of fever, headache or malaise) to anemia, we are planning a human iron absorption study in Benin. We will recruit adults with asymptomatic malaria infection. The iron absorption and utilization of the study subjects will be studied while infected, then they will be treated to clear their infections, and then iron absorption and utilization will be restudied. Iron absorption will be determined by incorporation of labeled iron into erythrocytes, 14 days after the administration of a test meal containing labeled iron (stable isotope technique). Subjects will be men and non-pregnant, non-breastfeeding women with a body weight < 65 kg and between the age of 18 - 30 years.

The results of this study will provide important information on the influence of malaria infections on iron absorption and utilization in humans. The study will provide insight into the potential necessity of malaria control to ensure iron bioavailability from foods in developing countries.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 y
* Body weight < 65 kg
* A positive malaria smear (asexual P. falciparum parasitemia > 500/μL blood) without clinical symptoms (fever or self-reported fever in last 7 days, headache, malaise)
* If female, not pregnant (tested by pregnancy test) and not breastfeeding
* No mineral and vitamin supplements two weeks before and during the study

Exclusion Criteria:

* Severe anemia (hemoglobin < 8.0 g/dl)
* Chronic medical illnesses
* Blood donation or transfusion in the last 6 months before study time
* Soil-transmitted helminth infections (positive Kato-Katz-Smear)
* Tuberculosis (TB): The potential presence of TB will be excluded by a short health questionnaire (cough? night sweats? weight loss? close relative with TB?). If this questionnaire raises the possibility that the subject may be at risk for TB, he/she will be referred to the local medical service

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2009-02; Primary Completion 2009-09 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zimmermann, Prof., MD, Principal Investigator — Human Nutrition Laboratory, Swiss Federal Institute of Technology
Locations (1):
- Hopital de zone de Natitingou, Natitingou, Natitingou, Benin

REFERENCES:
- [Derived] Cercamondi CI, Egli IM, Ahouandjinou E, Dossa R, Zeder C, Salami L, Tjalsma H, Wiegerinck E, Tanno T, Hurrell RF, Hounhouigan J, Zimmermann MB. Afebrile Plasmodium falciparum parasitemia decreases absorption of fortification iron but does not affect systemic iron utilization: a double stable-isotope study in young Beninese women. Am J Clin Nutr. 2010 Dec;92(6):1385-92. doi: 10.3945/ajcn.2010.30051. Epub 2010 Oct 6. PMID 20926522